CLINICAL TRIAL: NCT00435942
Title: Phase II Clinical Study of the Safety and Efficacy of the Relay Thoracic Stent-Graft in Patients With Thoracic Aortic Pathologies
Brief Title: Phase II Study of the Safety and Efficacy of the Relay Thoracic Stent-Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-0004-06; NCT00998491 (obsolete NCT alias)
Expanded Access: NCT01327742 (Approved for marketing)
Record Dates: First submitted 2007-02-14; First posted 2007-02-16 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-08

CONDITIONS: Thoracic Aortic Aneurysms; and Penetrating Atherosclerotic Ulcers
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Penetrating Atherosclerotic Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Endovascular Treatment arm to be implanted with Relay device
  Interventions: Device: Relay Thoracic Stent-Graft
- 2 (Active Comparator): Surgical Control, underwent open repair
  Interventions: Procedure: Open Repair

INTERVENTIONS:
Device: Relay Thoracic Stent-Graft — implant
  Arms: 1
Procedure: Open Repair — Open surgery
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Relay thoracic stent-graft system to treat thoracic aortic aneurysms. Efficacy will be evaluated by the device-related adverse event rate of endovascular repair (via Relay Thoracic Stent-Graft) through 1-year. Safety will be evaluated by comparing major adverse events through 1-year in subjects treated with the Relay Thoracic Stent-Graft to those who underwent surgical repair. Long term follow-up is conducted through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosed descending thoracic aortic aneurysms or penetrating atherosclerotic ulcers
* Subjects who are at least 18 years of age
* Subjects whose anatomy can accommodate the Relay device
* Subjects who consent to participate
* Subjects who agree to comply with follow-up schedule

Exclusion Criteria:

* Subjects with non-aneurysm lesions
* Subjects with less than 1 year life expectancy
* Subjects who are pregnant
* Subjects with medical conditions that would complicate the endovascular procedure or confound the results (e.g., Marfan's Syndrome, prior repair in the thoracic aorta, severe coronary artery disease, morbid obesity, etc.)
* Subjects participating in another investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-01; Primary Completion 2011-04 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Farber, MD, Principal Investigator — University of North Carolina
Locations (27):
- United States (27):
  - Arizona Heart Hospital, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California-San Francisco, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Rockford Memorial Hospital, Rockford, Illinois
  - Clarian Cardiovascular, Indianapolis, Indiana
  - Indiana Heart Hospial, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - The Mayo Clinic, Rochester, Minnesota
  - Albany Medical Center, Albany, New York
  - New York Presbyterian Hospital --Columbia/Cornell University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania/Penn Presbyterian, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Methodist Hospital, Houston, Texas
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Sentara Heart Hospital, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - Aurora St. Luke's Hospital, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects screened and enrolled at 29 sites in the United States
Groups:
- Relay Device Group: Endovascular Treatment arm
- Surgical Control Group: Open Surgical Repair arm
Period: Overall Study
Arm/Group | Relay Device Group | Surgical Control Group
Started | 120 | 60
Completed (97 patients) | 97 | 33
Not Completed | 23 | 27
Not completed — Death | 17 | 10
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 16
Not completed — Conversion to Open Repair | 1 | 0
Not completed — Technical Failure | 3 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relay Device Group | Surgical Control Group | Total
Number analyzed (Participants) | 120 | 60 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 12 | 33
  >=65 years | 99 | 48 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (11.02) | 70.0 (9.17) | 71.84 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 20 | 78
  Male | 62 | 40 | 102
Region of Enrollment [Number; unit: participants]
  United States | 120 | 60 | 180

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint: Freedom From Major Adverse Device Effects
Description: The primary effectiveness endpoint was freedom from major device-related adverse events [endoleak (Types I, III and IV), stent migration (> 10mm as compared to the 1 month visit), lumen occlusion, aneurysm rupture, and deployment failure/conversion to surgical repair] at 1 year post-procedure.
  The proportion of participants in the Effectiveness sample who were free from major device-related AEs at 1-year post-procedure was compared against a performance goal of 0.80 using a 1-sided z-test (normal approximation to the binomial) at an alpha level of 0.025. Rejection of the null hypothesis would provide evidence that this performance goal (proportion-free greater than 0.80) was met.
Time Frame: 1 year
Population: All subjects who underwent the Relay implant procedure (Intention to Treat)
Measure: Number; unit: participants
Arm/Group | Relay Device Group
Number analyzed (Participants) | 120
participants | 97
Statistical Analysis 1: Comparison: Relay Device Group; The proportion of subjects in the Effectiveness sample who were free from major device-related AEs at 1-year post-procedure was compared against a performance goal of 0.80 using a 1-sided z-test (normal approximation to the binomial) at an alpha level of 0.025. Rejection of the null hypothesis would provide evidence that this performance goal (proportion-free greater than 0.80) was met; Test type: Non-Inferiority or Equivalence — The proportion of subjects in the Effectiveness sample who were free from major device-related AEs at 1-year post-procedure was compared against a performance goal of 0.80 using a 1-sided z-test (normal approximation to the binomial) at an alpha level of 0.025. Rejection of the null hypothesis would provide evidence that this performance goal (proportion-free greater than 0.80) was met; p > 0.80, 1-sided z-test; 97.5% 1-sided confidence interval; Proportion free = 0.97, 97.5% CI 1-sided [lower limit .93]

2. Primary Outcome: Primary Safety Endpoint: Distribution of Major Adverse Events
Description: The primary safety endpoint was the distribution of participants experiencing at least 1 of the major adverse events (aneurysm-related mortality, stroke, paralysis/paraplegia, myocardial infarction, procedural bleeding, respiratory failure, renal failure, and wound healing complications) within 1 year post-procedure
Time Frame: 1 year
Population: The number of subjects who underwent the endovascular procedure or open surgical repair
Measure: Number; unit: participants
Arm/Group | Relay Device Group | Surgical Control Group
Number analyzed (Participants) | 120 | 60
participants | 27 | 51

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for 1 year per participant, up to Day 673.
Description: Adverse Events grouped by organ system
Arm/Group | Relay Device Group | Surgical Control Group
Serious Adverse Events (participants affected / at risk) | 68/120 | 45/60
Other Adverse Events (participants affected / at risk) | 97/120 | 58/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relay Device Group (N=120) | Surgical Control Group (N=60)
Bleeding events (Injury, poisoning and procedural complications) | 12 (13) | 33 (37)
Cardiac complications (Cardiac disorders) | 21 (32) | 12 (18)
Endoleak (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Hematology complications (Blood and lymphatic system disorders) | 6 (10) | 3 (3) — Includes anemia, coagulopathy, increased platelets
Neurological complications (Nervous system disorders) | 19 (22) | 8 (13) — Includes stroke, paraplegia, paraparesis
Pulmonary Complications (Respiratory, thoracic and mediastinal disorders) | 20 (28) | 20 (27)
Renal/genitourinary complications (Renal and urinary disorders) | 12 (15) | 6 (6)
Vascular complications (Vascular disorders) | 10 (12) | 5 (6) — Includes ruptures of untreated aneurysms, aortic dissecton
Vascular access complications (Vascular disorders) | 4 (5) | 0 (0) — includes access difficulty, iliac artery injury
General (General disorders) | 15 (19) | 7 (10) — includes a variety of event types (e.g., decreased nutritional intake, volume overload, etc.)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Digestive/gastrointestinal complications (Gastrointestinal disorders) | 7 (7) | 8 (9)
Dermatological complications (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Device malfunctions (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.8% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Relay Device Group (N=120) | Surgical Control Group (N=60)
Bleeding Events (Injury, poisoning and procedural complications) | 22 (26) | 25 (26) — Includes procedural bleeding and post-procedural bleeding
Cardiac complications (Cardiac disorders) | 35 (56) | 27 (36)
Endoleak (Injury, poisoning and procedural complications) | 14 (16) | 0 (0)
Hematology complications (Blood and lymphatic system disorders) | 28 (58) | 19 (26) — Includes anemia, coagulopathy, thrombocytopenia
Neurological complications (Nervous system disorders) | 39 (53) | 20 (22)
Pulmonary complications (Respiratory, thoracic and mediastinal disorders) | 30 (50) | 35 (66)
Renal/genitourinary complications (Renal and urinary disorders) | 24 (36) | 9 (14)
Vascular complications (Vascular disorders) | 9 (10) | 2 (2)
Vascular Access Complications (Vascular disorders) | 10 (10) | 0 (0)
General (General disorders) | 55 (127) | 31 (61)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Digestive/gastrointestinal complications (Gastrointestinal disorders) | 32 (51) | 14 (17)
Dermatological Complications (Skin and subcutaneous tissue disorders) | 21 (30) | 14 (20)
Device Malfunctions (Injury, poisoning and procedural complications) | 2 (5) | 0 (0)
Trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Localized pain (Injury, poisoning and procedural complications) | 23 (23) | 3 (3)
Hepatic complications (Hepatobiliary disorders) | 2 (2) | 0/0 (0)

LIMITATIONS AND CAVEATS:
Many subjects experienced more than one type of event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator must provide Bolton Medical with the proposed publication for review. Bolton Medical had 30 days to review and had discretion to make changes.